CLINICAL TRIAL: NCT03610568
Title: The Global Early Adolescent Study, Phase 2 | Kinshasa, Democratic Republic on the Congo
Brief Title: Global Early Adolescent Study - Kinshasa
Acronym: GEAS_KI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Save the Children (Other); Bill and Melinda Gates Foundation (Other); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7510
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Gender Relations; Reproductive Health
Keywords: Gender Norms; Gender-Based Violence; Mental Health; Sexual & Reproductive Health; Adolescent Health
MeSH Terms: conditions — Psychological Well-Being; Coitus

STUDY DESIGN:
Intervention Model Description: 1,400 adolescents were enrolled in the intervention group - 1,000 in-school and 400 out-of-school 1,400 adolescents were enrolled in the control group - 1,000 in-school and 400 out-of-school
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growing up GREAT! Intervention (Experimental)
  Interventions: Behavioral: Growing up GREAT! Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Growing up GREAT! Intervention — The Growing up GREAT! intervention is built around the socio-ecological model. For young adolescents, a suite of materials provides information and prompts discussion about puberty, gender equality, healthy relationships, violence, and other related themes during weekly club sessions. For parents, group sessions featuring six testimonial videos foster discussion around non-violent parenting, equal sharing of household tasks, and girls' education. Other materials for teachers, health workers, and community members complement the core toolkit materials.
  Arms: Growing up GREAT! Intervention

SUMMARY:
The Global Early Adolescent Study (GEAS) is the first international study exploring how gender norms evolve over time and inform a spectrum of adolescent health outcomes, including sexual and mental health, through the adolescent years. Institutional Review Board (IRB) oversight for all instrument development was provided for the first phase of the GEAS under IRB #00005684. The present study is in reference to the second, longitudinal phase of the GEAS. This phase, like the first, will be conducted in multiple international sites. However, because the longitudinal phase will likely be paired with different interventions or approaches in the partner sites, protocol details will vary and thus IRB approval will be sought for each site separately. The present application is for conducting Phase 2 of the Global Early Adolescent Study in Kinshasa, Democratic Republic of the Congo (DRC). In addition to conducting the study for "pure science" purposes, the GEAS will be used to evaluate the effectiveness of an intervention implemented by Save the Children.

DETAILED DESCRIPTION:
The Global Early Adolescent Study (GEAS) is the first international study exploring how gender norms evolve over time and inform a spectrum of adolescent health outcomes, including sexual and mental health, through the adolescent years. The first phase, consisting of formative research and the face validity and pilot testing of instruments among early adolescents 10-14 years of age across 15 countries, was completed in 2017.

The present study is for Phase 2 of the Global Early Adolescent Study in Kinshasa, Democratic Republic of the Congo (DRC), and covers both the intervention and control groups. The longitudinal phase explores how gender norms relate to health across the adolescent years, beginning with early adolescence (10-14 years old). The GEAS in Kinshasa has two sets of objectives:

1. To explore how perceptions of gender norms evolve across adolescence, the factors influencing these changes, and how perceptions of gender norms predict a spectrum of adolescent outcomes, and
2. Assess the impact of a gender norms transformative intervention developed and implemented by Save the Children.

The intervention, Growing Up GREAT (GUG), and evaluation components are part of a larger project, Passages, which is led by the Institute for Reproductive Health (IRH) at Georgetown University. The investigator's research partner is the Kinshasa School of Public Health (KSPH), which will implement the GEAS study. Through Passages, Johns Hopkins University (JHU) receives support primarily from USAID with additional support from the Bill and Melinda Gates Foundation as a sub-recipient of IRH. Save the Children is separately a sub-recipient of IRH. This funding supports 3 years of longitudinal research with both control and intervention groups for impact evaluation in Kinshasa.

In both an intervention and control group 1,400 young people ages 10-14 will be followed over a period of 3 years, participating in a total of 3 surveys. To gauge effectiveness of the intervention, the study will assess the following measurable primary and secondary study outcomes:

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 10-14 years of age
* Lives within the geographic boundaries of Kimbanseke or Masina
* Lives at home with a family (biological, adoptive, or foster)
* Attends a school selected for the study

INTERVENTION GROUP ONLY

* Has indicated interest in participation in the after-school component of the intervention
* Able to assent
* Has obtained informed consent from a parent or guardian to participate in the study

Exclusion Criteria:

* Not between the ages of 10-14
* Does not live within the geographic boundaries of Kimbanseke or Masina
* Is homeless or lives on the street
* Attends a school not selected for the study, or does not attend school

INTERVENTION GROUP ONLY

* Attends a school selected for the study but has not indicated interest in participation in the after-school component of the intervention
* Unable to assent
* Has not obtained informed consent from a parent or guardian to participate in the study

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2862 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Contraceptive use as assessed by self-reported use at last sex from the Global Early Adolescent Study Questionnaire | 3 years
  Change in contraceptive prevalence among sexually active adolescents
Exposure to gender-based violence in the past 6 months as assessed by self-report from the Global Early Adolescent Study Questionnaire | 1 year
  Change in reports of exposure to gender-based violence (GBV) at Wave II compared with baseline, sustained over subsequent waves of data collection.

SECONDARY OUTCOMES:
Gender-equitable attitudes and beliefs from the Global Early Adolescent Study Questionnaire | 3 years
  Shift in self-reported gender-equitable attitudes and beliefs

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Moreau, MD, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes